CLINICAL TRIAL: NCT00407212
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter, Dose-ranging, Efficacy and Safety Study of Three Doses of TCH346 (1mg, 5mg and 20mg Daily) in Patients With Early Parkinson's Disease
Brief Title: A Study of Three Doses of TCH346 in Patients With Early Parkinson's Disease to Evaluate Safety and Efficacy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCH346B103
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Parkinson's Disease
Keywords: early stage idiopathic Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — dibenzo(b,f)oxepin-10-ylmethyl-methyl-prop-2-ynyl-amine

INTERVENTIONS:
Drug: TCH346 (dibenz[b,f]oxepin-10-ylmethyl-prop-2-ynyl-amine, hydrogen maleate salt)

SUMMARY:
This study will investigate the effect of TCH346 compared to placebo in delaying the need for symptomatic treatment with dopaminergic agents

DETAILED DESCRIPTION:
This study will investigate the effect of TCH346 compared to placebo in delaying the need for symptomatic treatment with dopaminergic agents

ELIGIBILITY:
Inclusion Criteria:

* Male or female ,aged 30-80 years
* Clinical diagnosis of early stage idiopathic Parkinson's disease
* Experiencing two of the three following signs; bradykinesia, rigidity, and tremor
* Not currently taking any antiparkinson medication

Exclusion Criteria:

* A history of alcohol or drug abuse in the past year
* A diagnosis psychiatric illness
* Patients who currently are taking MAO inhibitors within 30 days of entering the study
* Patients who are hypersensitive to selegiline, MAO-B inhibitors, or tricyclic antidepressants

Additional inclusion/exclusion criteria may apply

Ages: 30 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2002-01; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Time to the need for symptomatic treatment with dopaminergic agents", defined as the number of days from the first dose of TCH346 study treatment to the date when it symptomatic treatment is required as determined by the investigator
Safety assessments as based on the frequency of adverse events and the number of laboratory values that fall outside of the ranges.

SECONDARY OUTCOMES:
Annual change rates for Unified Parkinsons Disease Rating Scalescore
Changes in UPDRS score after 4 weeks and after withdrawal of study treatment
Percentage of patients needing symptomatic treatment within 12 months

CONTACTS AND LOCATIONS:
Locations (45):
- United States (11):
  - Phoenix, Arizona
  - Berkley, California
  - Fountain Valley, California
  - Sunnyvale, California
  - New Haven, Connecticut
  - Chicago, Illinois
  - Southfield, Michigan
  - Great Falls, Montana
  - Columbus, Ohio
  - Pawtucket, Rhode Island
  - Houston, Texas
- Brazil (4):
  - Novartis Investigative Site, Belo Horizonte
  - Novartis Investigative Site, Curitiba
  - Novartis Investigative Site, Fortaleza
  - Novartis Investigative Site, São Paulo
- Canada (6):
  - Novartis Investigative Site, Caligary
  - Novartis Investigative Site, Hallifax
  - Novartis Investigative Site, Markham
  - Novartis Investigative Site, Montreal
  - Novartis Investigative Site, Vancouver
  - Novartis Investigative Site, Winnipeg
- France (5):
  - Novartis Investigative Site, Clermont
  - Marseille
  - Novartis Investigative Site, Paris
  - Saint-Herblain
  - Tours
- Germany (4):
  - Berlin
  - Bochum
  - Leipzig
  - Wiesbaden
- Italy (5):
  - Genova
  - Lido di Camaiore
  - Maples
  - Milan
  - Pescara
- Netherlands (6):
  - 's-Hertogenbosch
  - Amsterdam
  - Bedra
  - Biaricum
  - Dordrecht
  - Groningen
- Lisbon, Portugal
- United Kingdom (3):
  - Birmingham
  - Cambridge
  - Sheffield